CLINICAL TRIAL: NCT04432519
Title: Linear and Volumetric Analysis on the Effect of Customized Healing Abutments at Maxillary Immediate Implant Sites: a Prospective Randomized Clinical Trial
Brief Title: Multi-level Dimensional Changes at Immediate Implant Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Católica Portuguesa (Other)
Collaborators: Danilo Fernandes (Unknown)
Responsible Party: Principal Investigator, Tiago Borges, Professor, Universidade Católica Portuguesa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06.2019
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Dental Implant Failed

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group CA (Experimental): Customized healing abutment inserted in immediate implant placement.
  Interventions: Procedure: Immediate dental implant placement
- Group CM (Active Comparator): Resorbable Collagen Membrane for socket closure in immediate implant placement.
  Interventions: Procedure: Immediate dental implant placement

INTERVENTIONS:
Procedure: Immediate dental implant placement — Dental implant insertion in the same surgical stage of the tooth extraction, consisting in implant placement in the fresh socket.
  Other Names: Post extraction immediate implant placement

SUMMARY:
Studies evaluating the use of customized healing screws/abutments in immediate implant placement have been performed, aiming to assess possible advantages with the use of this treatment modality. Despite the existence of these investigations, there is a lack of information regarding a digital approach to evaluate in an objective manner soft and hard tissue dimensional changes at this treatment modality.

DETAILED DESCRIPTION:
Studies evaluating the use of customized healing screws/abutments have been performed aiming to assess possible advantages with the use of this treatment modality. Despite the existence of these investigations, there is a lack of information regarding a digital approach to evaluate in an objective manner soft and hard tissue dimensional changes.

The aim of this study is to perform a volumetric analysis evaluating peri-implant tissues dimensional changes on the effect of using customized healing abutments compared with the use of collagen matrices as socket sealing options in maxillary immediate implant placement.

The present study was designed as a prospective, randomized, controlled clinical trial with a parallel-group design, to document the response of using a customized healing abutment in maxillary immediate implants. Twenty-eight consecutive patients in need of a single implant restoration in the maxillary arch following tooth extraction were included in this study.

All patients were treated with cylindrical shape implants (OsseoSpeed EV™, AstraTech Implant System, Dentsply Implants, Möhndal, Sweden) with a narrow diameter internal connection platform following the surgical sequence protocol provided by the manufacturer. The implant was placed in a correct three-dimensional position, engaging the palatal and apical bone to achieve high primary stability. (Buser et al. 2004) After implant insertion, a gap of at least 2 mm between the inner cortical buccal bone plate and the implant surface was filled with DBBM material (Symbios®, Dentsply Implants, Möhndal, Sweden).

The two groups differ in the type of socket sealing. Control group fresh sockets were sealed with a resorbable collagen membrane (Mucograf Seal®, Geistlish Biomaterials, Wolhusen, Switzerland) stabilised with single interrupted 6/0 polyamide sutures (SeralonTM, Serag-Wiessner, Nalia, Germany), whereas test group received a healing abutment customized with a composite resin material allowing to close the socket without sutures.

Clinical examination and image acquisition Examination protocol and data collection consisted of four appointments: 1) T0 (flapless tooth extraction and implant insertion; 2) T1 (1-month follow-up after implant placement; 3) T2 (4-month follow-up after implant insertion) and 4) T3 (1-year postoperative follow-up). An intraoral scan of the upper arch (Cerec Omnicam®, Sirona Dental Systems GmbH, Bensheim, Germany) and a CBCT radiographic evaluation (Ortophos XG 3D®, Sirona Dental Systems GmbH, Bensheim, Germany) were performed followed by tooth extraction and implant placement (T0). At this point, two clinical parameters were assessed with a periodontal probe to the nearest millimetre: BID (distance between implant shoulder and the buccal bone plate) and KM (distance between the gingival groove and the mucogingival junction). Intraoral scans were completed post-implant placement at one month (T1), four months (T2) and twelve months (T3). In all follow-up appointments hygiene instructions were given to the patients and a periodontal care was executed when necessary.

Matching digital models All digital models were exported from the intraoral scanner in STL format. The T0 and T1, T0 and T2, and T0 and T3 STL files were overlapped and a strict alignment was made into one common coordinate system. A final alignment was done through the best fit alignment algorithm for a perfect match of digital models and executed with settings adjusted to the oral cavity.

After the superimposition of digital models, a colour map was created to quantitatively analyse the three-dimensional changes occurring in the surgical areas and adjacent tissues. Green areas correspond to the perfect alignment of the model. The variation between yellow and red represents variations of volumetric increase, whereas the variations between light blue and dark blue represent the variations of volumetric decrease. A region of interest (ROI) with 10 section planes, perpendicular to the coronal section of the tooth, was computed at buccal and palatal aspect (Figure 2). These sections were set at the most apical point of the gingival margin and ended 5 mm above it. Mesially and distally, a line passing through the interproximal area limited the region of interest. The same ROI was used in each patient, at the different comparison points. The intersection of these sections with the overlapping models allowed the linear changes to be obtained in each area. The Mean Buccal Change (MBC0-1, MBC0-2, and MBC0-3) and Mean Total Change (MTC0-1, MTC0-2 and MTC0-3) were calculated in millimetres (mm) to evaluate the changes that occurred in peri-implant contour (Figure 3).

Digital models superimposed in Geomagic Control X® were exported to Materialise Magics® for volumetric assessment. A volumetric ROI was manually selected with "Cut or Punch" function using interproximal areas as mesial and distal limits. All cuts were performed in the same way in all digital models so that all measurements were carried out in the same areas. ROI volume at T0 was computed for further comparison with consecutive volume variation values (Figure 4). The 3D-analysis was conducted with "Boolean" functions, which allowed researchers to obtain the volume variation in each time point from different variables like the Buccal Volume Variation (BVv0-1, BVv0-2, and BVv0-3) and Total Volume Variation (TVv0-1, TVv0-2, e TVv0-3), computed in cubic millimetres (mm3). To allow a direct comparison of different sites at different time points, relative percentages of these variables were calculated based on the ROI volume at T0 (Szathvary et al. 2015). All measurements were recorded to the nearest 0.01 mm.

Radiographic assessment The acquisition of radiographic images was performed with a volumetric dimension of 8 x 8 cm for 14s with the tomography acquisition protocol, with a voxel size of 0.1 mm in HD mode. The CBCT images were imported in a DICOM format to Mimics® software to perform the measurements. Buccal plate thickness (BT) was assessed for 3D radiographic analysis to evaluate the initial features of the alveolar bone. All measurements were obtained through coronal slice reconstructions, using an adjacent line to the sinus/nasal plate as a reference (Figure 5). BT was measured 1 mm above the coronal bone margin using a central slice, as well at the mesial and distal slices, ranging 1 mm from the central slice. Mean BT values were obtained as the average values of the three slices. One independent examiner who was not involved in the study executed all measurements.

Statistical analysis The outcome variables were presented as mean values, standard deviation, median and 95% confidence interval. Measurement time (T1, T2 and T3) was considered as a factor and the following as covariates: age, gender, KM height, location, implant length, BID and BT. The statistical analysis was performed using SPSS™ Statistical Package for the Social Sciences, version 21.0 (IBM Corporation, Armonk, NY, USA). The Mann-Whitney U-test was used to disclose differences for continuous non-paired variables. Moreover, the paired Wilcoxon test was used when the normal distribution of the groups was proved. A multiple linear regression model, using the stepwise forward method, was built to analyse the effect of the tested treatment in the main outcome variables throughout the study. All hypothesis tests were conducted at the 5% level of significance.

ELIGIBILITY:
Inclusion Criteria:

* patients with ≥18 years of age;
* patients who had a failing tooth and needed an implant placing therapy in the aesthetic zone (between 15-25);
* the failing tooth has adjacent and opposing natural teeth;
* sufficient mesial-distal and inter-occlusal space for placement of the implant and definitive restoration;
* had an intact socket wall previously to the extraction;
* had sufficient apical bone to place an immediate implant with minimum primary stability of 30 N/cm.

Exclusion Criteria:

* individuals diagnosed with periodontal disease;
* medical and general contraindications for the surgical procedure;
* heavy smokers (> 10 cigarettes/day); .an active infection at the implant site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Buccal volume variation (BVv) | Baseline (T0); 1 month (T1); 4 months (T2) and 12 months (T3)
  Variation of the alveolar volume at the buccal aspect. The 3D-analysis was conducted with "Boolean" functions, which allowed researchers to obtain the volume variation in each time point from different variables like the Buccal Volume Variation (BVv0-1, BVv0-2, and BVv0-3), computed in cubic millimetres (mm3) and To allow a direct comparison of different sites at different time points, relative percentages of these variables were calculated based on the ROI volume at T0.
Total volume variation (TVv) | Baseline (T0); 1 month (T1); 4 months (T2) and 12 months (T3)
  Variation of the alveolar volume at the buccal and palatal side. The 3D-analysis was conducted with "Boolean" functions, which allowed researchers to obtain the volume variation in each time point from different variables like the Total Volume Variation (TVv0-1, TVv0-2, e TVv0-3), computed in cubic millimetres (mm3) and To allow a direct comparison of different sites at different time points, relative percentages of these variables were calculated based on the ROI volume at T0

SECONDARY OUTCOMES:
Buccal wall thickness (BT) | baseline
  measurement of the facial bone wall. The acquisition of radiographic images was performed with a volumetric dimension of 8 x 8 cm for 14s with the XG 3D tomography acquisition protocol, with a voxel size of 0.1 mm in HD mode. BT was measured 1 mm above the coronal bone margin using a central slice, as well at the mesial and distal slices, ranging 1 mm from the central slice. Mean BT values were obtained as the average values of the three slices. Measurements were made in mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Católica Portuguesa /FMD, Viseu, Portugal